CLINICAL TRIAL: NCT00969579
Title: Characterizing Lone Parenting: A Multi-Institutional Pilot Study of the Perceptions of Support and Perceived Stress of Lone Parents of Children With Cancer
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090194; 09-M-0194
Record Dates: First submitted 2009-08-29; First posted 2009-09-01 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2018-03-08

CONDITIONS: Cancer
Keywords: Cancer; Psychosocial Stress; Parenting
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will describe the perceptions of support and distress outcomes of single/lone parents of a child with cancer.

Background:

* Parents and families of children with chronic illnesses have stressors, including financial stress, role strains, separations, and interruptions in daily routines and plans for the future. All of these experiences may lead directly and indirectly to parental stress.
* The number of families headed by single or lone parents is increasing. Little work has been done to better understand if the needs of parents who are providing care for a child on their own differ from parents who do not classify themselves as lone. Identifying parents who may need additional support within a pediatric oncology setting is very important so that appropriate support is provided.

Objectives:

- To better understand the social, emotional, and practical effects of lone parents on children with cancer.

Eligibility:

* All parents whose child has been diagnosed with cancer between 6 and 18 months before enrolling on the study.
* Participants must be able to speak and read English

Design:

* Parents will be asked to complete a questionnaire during one of their child s clinic or hospital visits.
* The questionnaire will ask about the parenting experience since the child was diagnosed with cancer. It will ask about the support the parent has received from family and friends since the diagnosis.
* The questionnaire will take approximately 20 minutes to complete.

DETAILED DESCRIPTION:
Background:

* Research examining the potential impact of childhood chronic illness on parents and families has delineated a myriad of stressors that parents may experience, including financial stress, role strains, separations, interruptions in daily routines and plans for the future, and general uncertainty regarding the child s prognosis.
* All of these possible experiences may lead directly and indirectly to anxiety, depression, posttraumatic-stress, hopelessness, and feelings of loss of control in parents and families.
* The number of families headed by single, or lone parents has increased significantly, with 3 in 10 children now living in single parent homes.
* It is not known whether distress is greater for parents who are lone parents.
* Lone-parent families earn on average only 55% of what married-parent families earn, and are four times more likely to live in poverty.
* It is unclear how lone parents trying to navigate the complex needs of maintaining a home, family, and a chronically ill child adapt to these challenges.
* It is also unclear how many parents who check single on a standardized forced choice questionnaire format consider themselves to be lone when it comes to the experience of caring for their child with cancer.

Objective:

<TAB>

* Aim 1: To define and characterize lone parents
* Aim 2: To describe perceptions of social support and how they relate to lone and non-lone parenting
* Aim 3: To identify distress outcomes in parents of children with cancer who identify themselves as being lone when it comes to the experience of caring for a child with cancer

Study Population:

English and Spanish speaking parents of a child (1through 17 years) with a malignancy, diagnosed 6-18 months before recruitment will be invited to participate in this study.

Design:

-This is a pilot, exploratory study designed to describe the perceptions of support and distress outcomes of single/lone parents of a child with cancer. Participants will be administered a Lone Parent Support Questionnaire designed for this study. The study will be completed in one visit (<30mins).

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Parents or primary guardians of children (ages 6 months through 17 years) with any malignancy whose child is 6-18 months post-diagnosis.
  2. Ability to give informed consent.
  3. English or Spanish speaking

EXCLUSION CRITERIA:

1. Severe psychological distress which - in the judgment of the Principal or Associate Investigators at each respective collection site- would compromise the participant s ability to understand the questionnaire or is likely to interfere with the study procedures or results.
2. Relapse of malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2009-08-06; Study Completion 2018-03-08

CONTACTS AND LOCATIONS:
Overall Officials: Maryland Pao, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (10):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Miller Children's Hospital, Long Beach, California
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University Of Mississippi Medical Center, Jackson, Mississippi
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Akron Children's Hospital, Akron, Ohio
  - Oklahoma State University, Stillwater, Oklahoma
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Barakat LP, Kazak AE, Meadows AT, Casey R, Meeske K, Stuber ML. Families surviving childhood cancer: a comparison of posttraumatic stress symptoms with families of healthy children. J Pediatr Psychol. 1997 Dec;22(6):843-59. doi: 10.1093/jpepsy/22.6.843. PMID 9494321
- [Background] Barrera M, D'Agostino NM, Gibson J, Gilbert T, Weksberg R, Malkin D. Predictors and mediators of psychological adjustment in mothers of children newly diagnosed with cancer. Psychooncology. 2004 Sep;13(9):630-41. doi: 10.1002/pon.765. PMID 15334531
- [Background] Brown RT, Wiener L, Kupst MJ, Brennan T, Behrman R, Compas BE, David Elkin T, Fairclough DL, Friebert S, Katz E, Kazak AE, Madan-Swain A, Mansfield N, Mullins LL, Noll R, Patenaude AF, Phipps S, Sahler OJ, Sourkes B, Zeltzer L. Single parents of children with chronic illness: an understudied phenomenon. J Pediatr Psychol. 2008 May;33(4):408-21. doi: 10.1093/jpepsy/jsm079. Epub 2007 Sep 29. PMID 17906331